CLINICAL TRIAL: NCT02049086
Title: Pain Management for Veterans Filing Compensation Claims
Acronym: SBIRT LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: R34AT008318-01 (NIH); R34AT008318-01 (NIH)
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Pain
Keywords: SBIRT; Screening; Brief Intervention; Referral to Treatment; Pain-Management; Veterans
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SBIRT-PM (Experimental): Screening, Brief Intervention and Referral to Treatment with Pain-Management advice (SBIRT-PM)
  Interventions: Behavioral: SBIRT-PM
- Pain Module Only (Active Comparator): The pain module of SBIRT-PM with no substance abuse focus (Pain Module Only)
  Interventions: Behavioral: Pain Module
- No Additional Referral (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: SBIRT-PM — Screening, Brief Intervention and Referral to Treatment with Pain-Management advice (SBIRT-PM)
  Arms: SBIRT-PM
Behavioral: Pain Module — The pain module of SBIRT-PM with no substance abuse focus (Pain Module Only)
  Arms: Pain Module Only

SUMMARY:
This proposal will develop and test an indicated prevention strategy, Screening, Brief Intervention and Referral to Treatment with Pain-Management advice (SBIRT-PM), in Veterans who have filed a claim for a (military) service-connected injury for which they have requested financial compensation. Although typically only an information-gathering, forensic-styled examination, the Compensation examination is a crucial point of entry to VA care. Objectives are:

1. To finalize the procedures, manual, and training materials of SBIRT-PM. The goals of this stage will be (1) optimizing SBIRT-PM's appeal to Veterans concerned about their musculoskeletal conditions and their Compensation claims; and (2) finalizing the counseling materials and procedures.
2. To conduct a randomized clinical trial comparing SBIRT-PM to a no referral arm and a pain module only arm.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of OEF/OIF/OND
* Scheduled exam for back, neck, knee, or shoulder. These four body parts were selected because they are classified as MSD by the VBA and are common causes of chronic non-cancer pain. Including other conditions (e.g. osteomyelitis, muscle injuries) would introduce more heterogeneity in illness course.
* Able to participate psychologically and physically, able to provide informed consent, complete assessments, and participate in study procedures.
* Self-reports peak pain of at least 2 on a numeric pain rating scale (0 "no pain" to 10 "worst pain imaginable" in the last 28 days in the joint that is the focus of the claim. This broad pain inclusion criterion may be narrowed after the Counseling Refinement Stage. Some Veterans apply for service connection for injuries that are not currently symptomatic, in case the injury recurs. This criterion will exclude these asymptomatic Veterans
* Risky substance use within the last 28 days, defined as one of the following:

  1. Risky alcohol use: i.e. >14 drinks/week or>4 drinks/occasion for men 65 or younger; >7 drinks/week or >3 drinks/occasion for women. A standard drink will be 14 grams of absolute alcohol, equivalent to 12 oz of beer, 5 oz of wine, or 1.5 oz of 80-proof liquor
  2. Self-reported use of an illicit drug in the preceding 28 days. Use of opioids or sedative hypnotics not prescribed to the Veteran will be considered illicit drug use.Medical marijuana is legal in Connecticut but is illegal federally. Use of medical marijuana puts someone at some risk for future misuse of cannabis or other drugs and therefore will be treated as an illicit drug.
  3. Misuse of prescribed opioid medications in the preceding 28 days. Two questions adapted from the CIDI for use in a NIDA Clinical Trials Network study, were modified to describe misuse of prescribed opioid medications: "How often have you taken your pain medications in larger amounts than prescribed or for a longer period than prescribed?" and "How often have you used your pain medicines to get high, to relax, or to make you feel more alert?"

Exclusion Criteria:

* Will not be able to attend the follow-up appointments.
* Attended VA or non-VA substance abuse treatment during the three months prior to randomization. Veterans who are receiving mental health treatment but indicate it is not addressing substance use will be enrolled.
* Physiological dependence on alcohol, illicit drugs, or non-prescribed opioids. People with more severe dependence have not benefited from SBIRT in prior studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Risky substance use | baseline
  A week will be defined as having had risky substance use if it had alcohol use at risky levels ( >14 drinks/week or 4 on an occasion for men or 7/week and >3/day for women), or illicit drug use. Weeks will be considered positive for illicit use if there is either a positive toxicology screen or self-reported use on that week.
Pain | baseline
  The primary pain outcome will be the pain severity score form the Brief Pain Inventory
Service Use | baseline
  Service use will be coded for each week as whether the Veteran attended any pain related, substance abuse and/or mental health treatment. Attendance at treatment during a week will be defined as having any service use data (VA or self-reported use of non-VA services) indicating use. The difference in probability of attendance over time will be compared across treatment groups. Use of non-VA services, and whether substance abuse was addressed during a counseling session will be self-reported.
Risky substance use | week 4
  A week will be defined as having had risky substance use if it had alcohol use at risky levels ( >14 drinks/week or 4 on an occasion for men or 7/week and >3/day for women), or illicit drug use. Weeks will be considered positive for illicit use if there is either a positive toxicology screen or self-reported use on that week.
Risky substance use | week 12
  A week will be defined as having had risky substance use if it had alcohol use at risky levels ( >14 drinks/week or 4 on an occasion for men or 7/week and >3/day for women), or illicit drug use. Weeks will be considered positive for illicit use if there is either a positive toxicology screen or self-reported use on that week.
Pain | week 4
  The primary pain outcome will be the pain severity score form the Brief Pain Inventory
Pain | week 12
  The primary pain outcome will be the pain severity score form the Brief Pain Inventory
Service Use | week 4
  Service use will be coded for each week as whether the Veteran attended any pain related, substance abuse and/or mental health treatment. Attendance at treatment during a week will be defined as having any service use data (VA or self-reported use of non-VA services) indicating use. The difference in probability of attendance over time will be compared across treatment groups. Use of non-VA services, and whether substance abuse was addressed during a counseling session will be self-reported.
Service Use | week 12
  Service use will be coded for each week as whether the Veteran attended any pain related, substance abuse and/or mental health treatment. Attendance at treatment during a week will be defined as having any service use data (VA or self-reported use of non-VA services) indicating use. The difference in probability of attendance over time will be compared across treatment groups. Use of non-VA services, and whether substance abuse was addressed during a counseling session will be self-reported.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System (VACHS), West Haven, Connecticut, United States

REFERENCES:
- [Derived] Rosen MI, Becker WC, Black AC, Martino S, Edens EL, Kerns RD. Brief Counseling for Veterans with Musculoskeletal Disorder, Risky Substance Use, and Service Connection Claims. Pain Med. 2019 Mar 1;20(3):528-542. doi: 10.1093/pm/pny071. PMID 29800338